CLINICAL TRIAL: NCT05102084
Title: The Effect of Listening to Music During CPAP on the Agitation Levels and Compliance With CPAP of Intensive Care Patients With COVID-19: A Randomized Controlled Trial
Brief Title: The Effect of Listening to Music During CPAP on the Agitation Levels and Compliance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SÜMEYYE BİLGİLİ (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, SÜMEYYE BİLGİLİ, Nursing Fundamentals Graduate Student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU-SBİLGİLİ_001
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; COVID-19 Acute Respiratory Distress Syndrome
Keywords: Covid-19; Cpap; Adapt; listen to music
MeSH Terms: conditions — COVID-19; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients listening to music during CPAP application
  Interventions: Device: Listening to music with a bluetooth headset to patients receiving CPAP support
- Control group (No Intervention): Patients not listening to music during CPAP application

INTERVENTIONS:
Device: Listening to music with a bluetooth headset to patients receiving CPAP support — Listening to music with a bluetooth headset during the CPAP application to the patients and checking the compatibility on the CPAP device.
  Arms: Experimental group

SUMMARY:
Aim: This study was conducted to determine the effect of listening to music during CPAP on the agitation levels of intensive care patients who underwent CPAP due to COVID-19 and their compliance with the treatment.

Study Design: This study is a prospective, randomized, controlled clinical trial. Seventy-six intensive care patients with COVID-19 were included in this study and assigned to the music and control groups via the block randomization method. The study was completed with 70 patients. In this study, the patients and outcome assessors were not blinded. The Richmond Agitation and Sedation Scale (RASS) level, respiratory rate, oxygen saturation (SpO2), and mask air leakage amount were the result criteria.

Results: The mean RASS score of the patients in the intervention group was 2.14±0.69 before CPAP, 1.63±064 at the 1st minute, 0.89±0.58 at the 15th minute, and 0.74±0.61 at the 30th minute. The mean RASS score of the patients in the control group was 2.06±0.53 before CPAP, 1.80±0.58 at the 1st minute, 1.43±0.60 at the 15th minute, and 1.46±0.61 at the 30th minute of CPAP. There was a statistically significant difference between the groups at the 15th and 30th minutes (t=-3.81, p < .001; t=-4.89, p < .001, respectively).

ELIGIBILITY:
Inclusion Criteria:

1. over 18 years old
2. Received CPAP treatment for 1 day in the intensive care unit,
3. Not hearing impaired,
4. No sedation treatment
5. Not diagnosed with a psychiatric illness,
6. Hemodynamically stable,
7. Not taking drugs (such as digoxin, adrenaline, dopamine) that affect blood pressure and pulse rate
8. Patients with a Glasgow Coma Scale score of 14 and above will be accepted.

Exclusion Criteria:

1. The patient's desire to leave the study
2. be under the age of 18
3. putting the patient on mechanical ventilation
4. have a hearing impairment
5. Receiving sedation therapy
6. diagnosed with psychiatric illness
7. Using drugs (such as digoxin, adrenaline, dopamine) that affect blood pressure and pulse rate
8. Patients with a Glasgow Coma Scale score below 14 will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in agitation level | 30 minutes
  The agitation levels of patients were monitored with the Richmond Agitation and Sedation Scale
Compliance with CPAP | 30 minutes
  Measure of respiratory rate, oxygen saturation,mask air leakage amount

SECONDARY OUTCOMES:
Variation of agitation and CPAP compliance with time | 30 minutes
  Measurements were made before CPAP, at 1st, 15th and 30th minutes of CPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Reva Balcı Akpınar, Prof. Dr, Principal Investigator — https://avesis.atauni.edu.tr/reva
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No